CLINICAL TRIAL: NCT05017610
Title: A Single Arm Pilot Study to Evaluate the Safety and Feasibility of Inducing a Hypothyroxinemic State in Patients With Recurrent Glioblastoma
Brief Title: Inducing a Hypothyroxinemic State in Patients With Recurrent Glioblastoma or Gliosarcoma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Per the PI-slow accrual
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey James Olson, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002497; NCI-2021-02249 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00002497; WINSHIP5264-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-07-28; First posted 2021-08-24 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Recurrent Glioblastoma; Recurrent Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Triiodothyronine; Lomustine; Methimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (methimazole, lomustine, liothyronine) (Experimental): See Outline in Detailed Description.
  Interventions: Drug: Liothyronine; Drug: Lomustine; Drug: Methimazole

INTERVENTIONS:
Drug: Liothyronine — Given PO
  Other Names: L-Triiodothyronine; Therapeutic T3; Triiodothyronine
Drug: Lomustine — Given PO
  Other Names: 1-(2-Chloroethyl)-3-cyclohexyl-1-nitrosourea; 1-Nitrosourea, 1-(2-chloroethyl)-3-cyclohexyl-; Belustin; Belustine; CCNU; Cecenu; CeeNU; Chloroethylcyclohexylnitrosourea; Citostal; Gleostine; Lomeblastin; Lomustinum; Lucostin; Lucostine; N-(2-Chloroethyl)-N''-cyclohexyl-N-nitrosourea; Prava; RB-1509; WR-139017
Drug: Methimazole — Given PO
  Other Names: Tapazole

SUMMARY:
This early phase I trial studies the safety and feasibility of inducing a hypothyroxinemic state in patients with glioblastoma or gliosarcoma that has come back (recurrent). This trial aims to see if giving a specific thyroid hormone, such as methimazole and liothyronine, is safe and could benefit cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and feasibility of inducing a hypothyroxinemic state in patients with recurrent glioblastoma.

SECONDARY OBJECTIVES:

I. To evaluate the anti-tumor activity of inducing hypothyroxinemic state by assessing progression-free survival (PFS) and overall survival (OS).

II. To evaluate the correlation of PFS and OS with thyroid hormone levels. III. To evaluate the correlation of overall response rate (ORR) with thyroid hormone levels.

IV. To evaluate the correlation of potential side effects with T3 levels or methimazole dose.

OUTLINE:

CATEGORY 1 (normal baseline thyroid function and no levothyroxine replacement): Patients receive methimazole orally (PO) daily and lomustine daily. Treatment with lomustine repeats every 6 weeks for up to 6 cycles or 12 months. Patients may receive liothyronine PO twice daily (BID) when thyroid-stimulating hormone (TSH) is above upper normal limit. Treatment continues in the absence of disease progression or unacceptable toxicity.

CATEGORY 2 (baseline primary hypothyroidism in patients taking levothyroxine): Patients receive liothyronine PO BID to maintain lower free T4 below lower limit of normal and TSH and free T3 in the normal range. At the time of cessation of exogenous T4, patients receive lomustine every 6 weeks for up to 6 cycles or 12 months. Treatment continues in the absence of disease progression or unacceptable toxicity.

CATEGORY 3 (secondary/tertiary hypothyroidism): Patients receive liothyronine PO BID to maintain lower free T4 below lower limit of normal and free T3 within normal range. At the time of cessation of exogenous T4, patients receive lomustine every 6 weeks for up to 6 cycles or 12 months. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 70%) within a 14-day window prior to randomization
* Patients must have histologically confirmed glioblastoma (or gliosarcoma) at first or second recurrence after initial standard, control or experimental, therapy that includes at least radiation therapy (RT) and temozolomide (TMZ)
* Evidence of progressive disease (PD) by modified response assessment in neuro-oncology criteria (using the post-chemoradiation time point as baseline), defined by any of the following:

  * >= 25% increase in sum of products of perpendicular diameters of measurable enhancing lesions, compared with the smallest tumor measurement obtained either at the post-chemoradiation baseline (if no decrease) or best response (on stable or increasing steroid dose).
  * Any new measurable (> 1 x 1 cm) enhancing lesions after the post-chemoradiation scan
* A total of at least 2 serial magnetic resonance imaging (MRI) scans documented at Screening including: 1) a scan at the time of suspected tumor progression; and 2) a scan prior to the time of progression. Patients must have progressed after standard of care treatment (it typically includes surgery, radiation and temozolomide). Pseudoprogression or radiation necrosis has been ruled out
* Hemoglobin >= 9.0 g/dl (no transfusions allowed within 7 days of cycle 1 day 1 to meet entry criteria) (within 14 days of starting treatment)
* Absolute neutrophil count (ANC) >= 1,500/mcL (after at least 7 days without growth factor support or transfusion) (within 14 days of starting treatment)
* Platelets >= 100,000/mcL (no transfusions allowed within 7 days of cycle 1 day 1 to meet entry criteria) (within 14 days of starting treatment)
* International normalized ratio (INR) =< 1.5 (within 14 days of starting treatment)
* Partial thromboplastin time (PTT) < 1.5 x upper limits of normal (ULN) (within 14 days of starting treatment)
* Total bilirubin =< 1.5 times the institutional upper limit of normal (ULN) (within 14 days of starting treatment)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.0 times the ULN (within 14 days of starting treatment)
* High amylase or lipase above upper normal limit (UNL) (within 14 days of starting treatment)
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x ULN. Creatinine clearance should be calculated per institutional standard (within 14 days of starting treatment)
* Electrocardiogram corrected QT interval by Fridericia's formula (QTcF) < 450 ms (within 14 days of starting treatment)
* Clinically significant toxic effect(s) of the most recent prior anti-cancer therapy must be grade 1 or resolved (except alopecia)
* A minimum time of 28 days elapsed from the administration of any prior cytotoxic agents
* Have undergone recent surgery for recurrent or progressive brain tumor are eligible provided that:

  * Prior to surgery there was imaging evidence of measurable progressive disease (PD) as described above.
  * Craniotomy or intracranial biopsy site must be adequately healed and free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of randomization.
  * Initiation of study treatment is at least 14 days from prior surgery/biopsy
* Availability of tumor tissue representative of glioblastoma (GBM) from initial definitive surgery and/or, recurrent surgery, if performed
* Female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study administration. A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions. Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* Patients who received temozolomide within 28 days prior to starting first cycle under this study
* Optune device is not allowed
* Patients who received prior lomustine, carmustine wafers, bevacizumab or any other anti-angiogenic agent
* Dexamethasone at time of study entry is not allowed. After a stable dose of methimazole and T3 is reached, dexamethasone can be used with a dose determined by treating physician
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Computed tomography (CT) scan with contrast within 6 weeks from enrollment as it may influence thyroid tests due to the iodine content
* History of cardiac arrhythmias (in particular, sinus bradycardia, atrial fibrillation or flutter, atrioventricular [AV] block, prolonged QTc, ventricular arrythmias, pacemaker, or implantable cardiac defibrillator).). Significant cardiovascular disease (eg, myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 6 months prior to start of study therapy; angina requiring therapy; symptomatic peripheral vascular disease; left ventricular ejection fraction less than or equal to 35%;New York Heart Association class 3 or 4 congestive heart failure; or uncontrolled grade >= 3 hypertension (diastolic blood pressure >= 100 mmHg or systolic blood pressure >= 160 mmHg) despite antihypertensive therapy, or use of amiodarone within the last 6 months.
* Uncontrolled type 2 diabetes mellitus (T2DM) (HbA1C greater than 8%) or a history of frequent hypoglycemia, or significantly uncontrolled hyperglycemia
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects of the study drugs. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study drugs breastfeeding should be discontinued if the mother will be on treatment
* Early disease progression prior to 3 months (12 weeks) from the completion of RT-TMZ, unless histologically proven to be recurrent GBM
* Had more than 2 prior lines for chemotherapy administration. NOTE: In the 1st line adjuvant setting, combination of TMZ with an experimental agent, is considered one line of chemotherapy
* Any prior treatment with an intracerebral agent
* Receiving additional, concurrent, active therapy for GBM outside of the trial
* Extensive leptomeningeal disease and defined by the principal investigator (PI)
* History of allergy or hypersensitivity to any of the study treatments or any of their excipient
* Unable or unwilling to undergo brain MRI scans with gadolinium
* History of another malignancy in the previous 2 years, with a disease-free interval of < 2 years. Participant with prior history of in situ cancer or basal or squamous cell skin cancer are eligible
* Serious, non-healing wound, ulcer, bone fracture, or abscess
* Any cerebrovascular accident (including transient ischemic attacks) within the last 6 months prior to initiation of study treatment
* Any hemorrhage or bleeding event that is >= grade 3 based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), grade 2 intracranial hemorrhage, or persistent thrombotic/embolic event within 4 weeks prior to the start of study medication
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or symptomatic pleural effusion
* Active, known or systemic suspected autoimmune disease, including systemic lupus erythematosus, scleroderma, polyarteritis nodose, or auto-immune hepatitis
* Known history of hepatitis B, human immunodeficiency virus (HIV), or active hepatitis C infection requiring treatment with antiviral therapy
* History of bleeding diathesis (irrespective of severity)
* History of agranulocytosis
* History of pancreatitis
* Uncontrolled psychiatric illness or any condition that could make the subject noncompliant with the study procedures and/or study requirements
* Participant has not been on a stable dose of anticoagulants for at least 2 weeks before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to study completion, an average of 2 years
  Descriptive statistics (e.g., frequency and percentage) for each adverse event/severe adverse event will be tabulated by association and grade.

SECONDARY OUTCOMES:
Overall response rate | Up to study completion, an average of 2 years
  Will be assessed by Response Assessment in Neuro-Oncology Criteria. Will be summarized with the 2-sided 95% confidence interval using the Clopper-Pearson method.
Progression free survival | Up to study completion, an average of 2 years
  Kaplan-Meier methods will be used to estimate median survival time or time-specific survival rate with a 95% confidence interval.
Overall survival | Up to study completion, an average of 2 years
  Kaplan-Meier methods will be used to estimate median survival time or time-specific survival rate with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Olson, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute

IPD SHARING:
Plan to Share IPD: No